CLINICAL TRIAL: NCT04986202
Title: A Randomised, Double-blind, Placebo-controlled, Multi-center Sequential Phase 2b and Phase 3 Study to Evaluate the Efficacy and Safety of AZD4831 Administered for Up to 48 Weeks in Participants With Heart Failure With Left Ventricular Ejection Fraction > 40%
Brief Title: Study to Evaluate the Efficacy and Safety of AZD4831 in Participants With Heart Failure With Left Ventricular Ejection Fraction > 40%
Acronym: ENDEAVOR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D6580C00010; 2020-005844-47 (EudraCT Number)
Record Dates: First submitted 2021-06-18; First posted 2021-08-02 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Heart failure; Heart failure with preserved ejection fraction; HFpEF
MeSH Terms: conditions — Heart Failure | interventions — AZD4831

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A 2.5 mg (Experimental): AZD4831 2.5 mg
  Interventions: Drug: AZD4831
- Part A 5 mg (Experimental): AZD4831 5 mg
  Interventions: Drug: AZD4831
- Part A Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- Part B Dose based on Part A (Experimental): AZD4831 Dose based on Part A
  Interventions: Drug: AZD4831
- Part B Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AZD4831 — AZD4831
  Arms: Part A 2.5 mg; Part A 5 mg; Part B Dose based on Part A
Other: Placebo — Placebo
  Arms: Part A Placebo; Part B Placebo

SUMMARY:
This is a randomised, double-blind, placebo-controlled, multi-center sequential phase 2b and Phase 3 study to evaluate the efficacy and safety of AZD4831 administered for up to 48 Weeks in participants with heart failure with left ventricular ejection fraction > 40%. The study will consist of 2 separate parts, Part A and Part B, approximately 660 participants will be randomised in Part A, 820 in Part B.

ELIGIBILITY:
Inclusion Criteria:

Part A

1. ≥ 40 to ≤ 85 years of age, at the time of signing the informed consent.
2. Documented stable symptomatic HF (New York Heart Association Class II-IV) for at least 1 month at Screening (Visit 1) (transient HF in the setting of an MI does not qualify), with a medical history of typical symptoms of HF and receiving optimal therapy for HF as determined by the health-care physician.
3. LVEF > 40% at Screening (Visit 1). All participants will undergo a local echocardiogram at the Screening (Visit 1) with central reading to confirm the LVEF > 40% eligibility criteria before randomisation.
4. 6MWD ≥ 30 meters and ≤ 400 meters at Screening (Visit 1) and Randomisation (Visit 3). Difference in 6MWD between Screening and Randomisation must be < 50 meters.
5. KCCQ-TSS ≤ 90 points at Screening (Visit 1) and Randomisation (Visit 3)
6. NT-proBNP ≥ 250 pg/mL (sinus rhythm) or ≥ 500 pg/mL (atrial fibrillation/flutter) at Screening (Visit 1) for patients with BMI ≤30 kg/m2.

NT-proBNP ≥ 200 pg/mL (sinus rhythm) or ≥ 400 pg/mL (atrial fibrillation/flutter) at Screening (Visit 1) for patients with BMI > 30 kg/m2.

The ECG performed at Screening should be used for heart rhythm evaluation.

7.At least one of the following:

1. Structural heart disease, ie, LA enlargement and/or left ventricular hypertrophy at the echocardiogram performed at Screening (Visit 1). Left atrial enlargement is defined by at least 1 of the following: LA width (diameter) ≥ 3.8 cm or LA length ≥ 5.0 cm, or LA area ≥ 20 cm2 or LA volume ≥ 55 mL or LAVI > 34 mL/m2. Left ventricular hypertrophy is defined by septal thickness or posterior wall thickness ≥ 1.1 cm or LVMI > 95 g/m2 in women and > 115 g/m2 in men.
2. Spectral tissue Doppler echocardiography - E/e' ratio (average of septal and lateral) ≥ 13 at rest at the echocardiogram performed at Screening (Visit 1).
3. Indirectly estimated elevation of PASP by TRmax velocity > 2.8 m/s (280 cm/s) (PASP > 35 mmHg) at the echocardiogram performed at Screening (Visit 1) OR directly measured pulmonary capillary wedge pressure > 15 mmHg at rest within the past 12 months or > 25 mmHg at exercise documented by right heart catheterisation within 12 months prior to Screening (Visit 1).
4. HF decompensation within 6 months before Randomisation (Visit 3), defined as hospitalisation for HF or IV diuretic treatment for HF during an urgent, unscheduled visit without hospitalisation.

   8.Body mass index ≥ 18.0 kg/m2 and ≤ 45.0 kg/m2

   9.Male or female of non-childbearing potential.

   Part B
   1. Participant must be ≥ 40 to ≤ 85 years of age, at the time of signing the informed consent.
   2. Documented diagnosis of symptomatic HF (NYHA class II-IV) at Screening (Visit 1), and a medical history of typical symptoms/signs of heart failure ≥ 6 weeks before Screening (Visit 1), and receiving optimal therapy for HF as determined by the health-care physician, with at least intermittent need for diuretic treatment.
   3. LVEF >40% and evidence of structural heart disease (ie, left ventricular hypertrophy or

      left atrial enlargement [defined by at least one of the following:LA enlargement and/or left ventricular hypertrophy at the echocardiogram

      performed at Screening (Visit 1). Left atrial enlargement is defined by at least 1 of the following: LA width

      (diameter) ≥ 3.8 cm or LA length ≥ 5.0 cm, or LA area ≥ 20 cm2 or LA volume ≥ 55 mL or LAVI > 34

      mL/m2. Left ventricular hypertrophy is defined by septal thickness or posterior wall thickness ≥ 1.1 cm or

      LVMI > 95 g/m2 in women and > 115 g/m2 in men.]) documented by the most recent echocardiogram, or cardiac

      magnetic resonance imaging within the last 12 months prior to Screening (Visit 1). If no

      echocardiogram is available, it can be performed at Screening (Visit 1).
   4. 6MWD ≥ 30 meters and ≤ 400 meters at Screening (Visit 1) and Randomisation (Visit 2). Difference in 6MWD between Screening and Randomisation must be < 50 meters
   5. KCCQ-TSS ≤ 90 points at Screening (Visit 1) and Randomisation (Visit 2).
   6. NT-proBNP ≥ 250 pg/mL (sinus rhythm) or ≥ 500 pg/mL (atrial fibrillation/flutter) at Screening (Visit 1) for patients with BMI ≤ 30 kg/m2. NT-proBNP ≥ 200 pg/mL (sinus rhythm) or ≥ 400 pg/mL (atrial fibrillation/flutter) at Screening (Visit 1) for patients with BMI > 30 kg/m2. The ECG performed at Screening should be used for heart rhythm evaluation
   7. Body mass index ≥ 18.0 kg/m2 and ≤ 45.0 kg/m2
   8. Male or female of non-childbearing potential.

   Exclusion Criteria:

   Part A

   1 eGFR < 30 mL/min/1.73m2 (Chronic Kidney Disease-Epidemiology Collaboration formula) at Screening (Visit 1).

   2. Systolic blood pressure < 90 mmHg or ≥ 160 mmHg if not on treatment with ≥ 3 blood pressure lowering medications or ≥ 180 mmHg irrespective of treatments at Randomisation

   3. Heart rate > 110 bpm or < 50 bpm at Randomisation

   4. Life expectancy < 3 years due to other reasons than cardiovascular disease.

   5. History or ongoing allergy/hypersensitivity reactions to drugs (including but not limited to rash, angioedema, acute urticaria).

   6. Presence of any disease or condition rather than HF constituting the main reason for limiting the ability to exercise/reduced exercise capacity.

   7. Current decompensated HF and/or NT-proBNP > 5000 pg/mL at Screening (Visit 1)

   8. Documented history of ejection fraction ≤ 40%.i.e. HF with recovered ejection fraction. Transient ejection fraction decrease e.g. in the setting of an MI does not apply

   9. Any planned cardiovascular procedure (eg, coronary revascularisation, ablation of atrial fibrillation/flutter, valve repair/replacement, aortic aneurysm surgery, etc).

   10. Any cardiac event (eg, myocardial infarction, unstable angina), coronary revascularisation (percutaneous coronary intervention or coronary artery bypass grafting), ablation of atrial fibrillation/flutter, valve repair/replacement, implantation of a cardiac resynchronisation therapy device within 12 weeks prior to Screening (Visit 1) or between Screening and Randomisation. Patients who underwent a successful atrial fibrillation/flutter cardioversion, can be enrolled in the study after 4 weeks.

   14. Hb < 110 g/L (male) and < 100 g/L (female) or iron-deficiency with/without anaemia requiring ongoing or planned IV iron treatment.

   15. Participants with hyperthyroidism, uncontrolled hypothyroidism (including but not limited to TSH ≥10 mIU/mL), or any clinically significant thyroid disease as judged by the investigator.

   18. ALT or AST ≥ 2 × ULN at Screening (Visit 1).

   19. Pulmonary arterial hypertension, chronic pulmonary embolism, severe pulmonary disease including COPD (ie, requiring home oxygen, chronic nebulizer therapy or chronic oral steroid therapy, or hospitalization for exacerbation of COPD requiring ventilatory support within 12 months prior to Screening (Visit 1).

   20. Any active infection requiring oral, intravenous or intramuscular treatment at Screening (Visit 1) and/or at Randomisation.

   23 Any signs or confirmation of COVID-19 infection:
   * Suspected (as judged by PI) or confirmed COVID-19 within the last 2 weeks prior to Screening (Visit 1) or at Randomisation.
   * Hospitalisation for COVID-19 within the last 12 weeks prior to Screening (Visit 1).

     24. Any concomitant medications known to be a potent CYP3A4 inducers or inhibitors, eg, itraconazole, rifampicin, clarithromycin, or propylthiouracil

     29. Previous enrolment and randomisation in the present study. (Participants who where screened and screen failed and not randomised in Part A can be screened for possible entry to Part B).

   All exclusion criteria in Part A are applicable to Part B with the following exceptions:

   Exclusion criteria 4; 19

   Exclusion Criteria specific for Part B only [criteria numeration for Part B]

   4. Life expectancy < 2 years due to other reasons than cardiovascular disease.

   11. HF due to any of the following: known infiltrative cardiomyopathy (eg, amyloid, sarcoid, lymphoma, endomyocardial fibrosis), active myocarditis, constrictive pericarditis, cardiac tamponade, known genetic hypertrophic cardiomyopathy or obstructive hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy/dysplasia (ARVC/D), or uncorrected primary valvular disease.

   18. Primary pulmonary hypertension, chronic pulmonary embolism, severe pulmonary disease including COPD (ie, requiring home oxygen, chronic nebulizer therapy or chronic oral steroid therapy, or hospitalization for exacerbation of COPD requiring ventilatory support within 12 months prior to Screening [Visit 1]).

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 711 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (146):
- United States (21):
  - Research Site, Alexander City, Alabama
  - Research Site, Little Rock, Arkansas
  - Research Site, Sacramento, California
  - Research Site, Miami, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Ocala, Florida
  - Research Site, Evanston, Illinois
  - Research Site, Hazel Crest, Illinois
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, St Louis, Missouri
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Rosedale, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Pinehurst, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Knoxville, Tennessee
  - Research Site, Tullahoma, Tennessee
  - Research Site, Norfolk, Virginia
- Australia (4):
  - Research Site, Bedford Park
  - Research Site, Chermside
  - Research Site, Concord
  - Research Site, Frankston
- Belgium (7):
  - Research Site, Aalst
  - Research Site, Dendermonde
  - Research Site, Hasselt
  - Research Site, Huy
  - Research Site, Kortrijk
  - Research Site, Leuven
  - Research Site, Roeselare
- Brazil (9):
  - Research Site, Brasília
  - Research Site, Campina Grande do Sul
  - Research Site, Campinas
  - Research Site, Canoas
  - Research Site, Curitiba
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Bulgaria (5):
  - Research Site, Blagoevgrad
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
- Canada (8):
  - Research Site, Guelph, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, North York, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Trois-Rivières, Quebec
- Czechia (9):
  - Research Site, Brno
  - Research Site, Broumov
  - Research Site, Jaroměř
  - Research Site, Kolín
  - Research Site, Louny
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Příbram
  - Research Site, Zlín
- Denmark (7):
  - Research Site, Århus N
  - Research Site, Copenhagen
  - Research Site, Copenhagen O
  - Research Site, Hvidovre
  - Research Site, København NV
  - Research Site, Roskilde
  - Research Site, Viborg
- France (13):
  - Research Site, Bayonne
  - Research Site, Dijon
  - Research Site, La Tronche
  - Research Site, Le Coudray
  - Research Site, Montauban
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Rennes
  - Research Site, Saint-Brieuc
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Tourcoing
- Hungary (3):
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Nyíregyháza
- Japan (20):
  - Research Site, Fukui-shi
  - Research Site, Higashiohmi-shi
  - Research Site, Iwakuni-shi
  - Research Site, Kanazawa
  - Research Site, Kasugai-shi
  - Research Site, Kishiwada-shi
  - Research Site, Kure-shi
  - Research Site, Kyoto
  - Research Site, Matsumoto-shi
  - Research Site, Minamiku
  - Research Site, Nagano
  - Research Site, Naha
  - Research Site, Otaru-shi
  - Research Site, Ōita
  - Research Site, Ōmihachiman
  - Research Site, Sagamihara-shi
  - Research Site, Toshima-ku
  - Research Site, Ueda-shi
  - Research Site, Uwajima-shi
  - Research Site, Yokohama
- Netherlands (5):
  - Research Site, 's-Hertogenbosch
  - Research Site, Amsterdam
  - Research Site, Deventer
  - Research Site, Heerlen
  - Research Site, The Hague
- Poland (9):
  - Research Site, Bydgoszcz
  - Research Site, Lublin
  - Research Site, Rzeszów
  - Research Site, Skierniewice
  - Research Site, Tarnów
  - Research Site, Tczew
  - Research Site, Tychy
  - Research Site, Warsaw
  - Research Site, Wołomin
- Russia (7):
  - Research Site, Aramil
  - Research Site, Kemerovo
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Perm
  - Research Site, Saint Petersburg
  - Research Site, Tver'
- Slovakia (6):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Brezno
  - Research Site, Košice
  - Research Site, Nitra
  - Research Site, Prešov
- Sweden (6):
  - Research Site, Gothenburg
  - Research Site, Jönköping
  - Research Site, Lund
  - Research Site, Norrköping
  - Research Site, Örebro
  - Research Site, Stockholm
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Turkey (Türkiye) (2):
  - Research Site, Eskişehir
  - Research Site, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Lund LH, Lam CSP, Pizzato PE, Gabrielsen A, Michaelsson E, Nelander K, Ericsson H, Holden J, Folkvaljon F, Mattsson A, Collen A, Aurell M, Whatling C, Baldus S, Drelich G, Goudev A, Merkely B, Bergh N, Shah SJ. Rationale and design of ENDEAVOR: A sequential phase 2b-3 randomized clinical trial to evaluate the effect of myeloperoxidase inhibition on symptoms and exercise capacity in heart failure with preserved or mildly reduced ejection fraction. Eur J Heart Fail. 2023 Sep;25(9):1696-1707. doi: 10.1002/ejhf.2977. Epub 2023 Aug 22. PMID 37470101
- See also: Redacted_CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6580C00010&attachmentIdentifier=d0341baa-e973-48d0-95d4-91c806b29fca&fileName=D6580C00010_Redacted_CSP.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6580C00010&attachmentIdentifier=ac832783-a7d5-46b3-8823-8d5a77d1fa45&fileName=D6580C00010-Redacted_CSR_synopsis.pdf&versionIdentifier=
- See also: D6580C00010_Redacted_SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6580C00010&attachmentIdentifier=c7691e40-e2a4-4c14-826f-c6b7fe018451&fileName=D6580C00010_Redacted_SAP.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 142 study centres in 18 countries randomised participants.
Pre-assignment Details: Part B of the study was never started, results are only presented for Part A of the study.
  The discrepancy between the number of randomised participants and the number of participants in the full analysis set and the safety analysis set is because only randomized participants who have taken at least one dose of the investigational product (IP) were included in the analysis sets.
Groups:
- AZD4831 2.5 mg: Once-daily oral dosing of AZD4831 2.5 mg
- AZD4831 5 mg: Once-daily oral dosing of AZD4831 5 mg
- Placebo: Once-daily oral dosing of placebo
Period: Overall Study
Arm/Group | AZD4831 2.5 mg | AZD4831 5 mg | Placebo
Started (Participants randomised) | 235 | 240 | 236
Completed (Participants completed study) | 218 | 234 | 220
Not Completed | 17 | 6 | 16
Not completed — Death | 10 | 3 | 10
Not completed — Physician Decision | 3 | 1 | 2
Not completed — Withdrawal by Subject | 4 | 2 | 4

BASELINE CHARACTERISTICS:
Population: All participants who have been randomised to study treatment and who have received at least one dose of investigational product were included irrespective of their protocol adherence and continued participation in the study and with non-missing data at baseline and the analysis timepoint. Participants were analysed according to their randomised study medication assignment, irrespective of the treatment actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD4831 2.5 mg | AZD4831 5 mg | Placebo | Total
Number analyzed (Participants) | 234 | 240 | 235 | 709
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.5 (7.3) | 72.1 (7.1) | 72.5 (7.8) | 72.4 (7.4)
Age, Customized [Number; unit: Participants]
  < 65 Years | 34 | 42 | 30 | 106
  65 - 75 Years | 120 | 108 | 115 | 343
  > 75 Years | 80 | 90 | 90 | 260
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 119 | 96 | 322
  Male | 127 | 121 | 139 | 387
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 16 | 14 | 21 | 51
  Not Hispanic or Latino | 218 | 226 | 214 | 658
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 35 | 36 | 36 | 107
  Black or African American | 5 | 10 | 6 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 193 | 194 | 192 | 579
  Other | 1 | 0 | 1 | 2
  Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  Australia | 1 | 1 | 1 | 3
  Belgium | 3 | 3 | 3 | 9
  Brazil | 13 | 14 | 15 | 42
  Bulgaria | 33 | 32 | 31 | 96
  Canada | 8 | 8 | 6 | 22
  Czech Republic | 23 | 22 | 22 | 67
  Denmark | 8 | 9 | 8 | 25
  France | 6 | 7 | 6 | 19
  Hungary | 18 | 19 | 19 | 56
  Japan | 25 | 25 | 25 | 75
  Netherlands | 4 | 5 | 5 | 14
  Poland | 22 | 23 | 24 | 69
  Russian Federation | 5 | 5 | 5 | 15
  Slovakia | 25 | 26 | 25 | 76
  Sweden | 12 | 12 | 13 | 37
  Taiwan | 10 | 10 | 10 | 30
  Turkey | 1 | 2 | 1 | 4
  United States of America | 17 | 17 | 16 | 50

OUTCOME MEASURES:

1. Primary Outcome: Kansas City Cardiomyopathy Questionnaire -Total Symptom Score
Description: Kansas City Cardiomyopathy Questionnaire -Total Symptom Score change from baseline at 16 weeks compared with placebo Part A. The score ranges from 0 to 100, where a higher score represents a better patient outcome
Time Frame: Baseline - 16 weeks
Population: All participants who have been randomised to study treatment and who have received at least one dose of investigational product are included irrespective of their protocol adherence and continued participation in the study and with non-missing data at baseline and the analysis timepoint. Participants were analysed according to their randomised study medication assignment, irrespective of the treatment actually received.
Measure: Least Squares Mean (95% Confidence Interval); unit: Points
Arm/Group | AZD4831 2.5 mg | AZD4831 5 mg | Placebo
Number analyzed (Participants) | 211 | 221 | 220
Points | 10.70 [8.58 to 12.82] | 9.81 [7.73 to 11.90] | 11.62 [9.54 to 13.71]
Statistical Analysis 1: Comparison: AZD4831 2.5 mg; Test type: Superiority; p = 0.537, ANCOVA — Two-sided test; Treatment group, neutrophil count stratification factor and the baseline value are included in the model as explanatory variables; Mean Difference (Final Values) = -0.92, 95% CI 2-sided [-3.86 to 2.02] — Difference in adjusted mean change from baseline between AZD4831 and placebo
Statistical Analysis 2: Comparison: AZD4831 5 mg; Test type: Superiority; p = 0.221, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.81, 95% CI 2-sided [-4.71 to 1.09] — Difference in adjusted mean change from baseline between AZD4831 and placebo

2. Primary Outcome: Six Minute Walk Distance
Description: Six Minute Walk Distance change from baseline at 16 weeks compared with placebo Part A
Time Frame: Baseline - 16 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Meters
Arm/Group | AZD4831 2.5 mg | AZD4831 5 mg | Placebo
Number analyzed (Participants) | 210 | 223 | 223
Meters | 15.3 [9.4 to 21.2] | 18.2 [12.4 to 23.9] | 12.9 [7.2 to 18.7]
Statistical Analysis 1: Comparison: AZD4831 2.5 mg vs Placebo; Test type: Superiority; p = 0.559, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [-5.7 to 10.5] — Difference in adjusted mean change from baseline between AZD4831 and placebo
Statistical Analysis 2: Comparison: AZD4831 5 mg vs Placebo; Test type: Superiority; p = 0.195, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 5.3, 95% CI 2-sided [-2.7 to 13.3] — Difference in adjusted mean change from baseline between AZD4831 and placebo

3. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire-Total Symptom Score
Description: Kansas City Cardiomyopathy Questionnaire -Total Symptom Score change from baseline at 24 and 48 weeks compared with placebo Part A. The score ranges from 0 to 100, where a higher score represents a better patient outcome.
Time Frame: Baseline - 24 and 48 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Points
Arm/Group | AZD4831 2.5 mg | AZD4831 5 mg | Placebo
Number analyzed (Participants) | 234 | 240 | 235
Points
  Kansas City Cardiomyopathy Questionnaire -Total Symptom Score change from baseline at 24 weeks: number analyzed (Participants) | 208 | 225 | 210
  Kansas City Cardiomyopathy Questionnaire -Total Symptom Score change from baseline at 24 weeks | 11.13 [8.94 to 13.32] | 11.92 [9.80 to 14.03] | 12.78 [10.59 to 14.97]
  Kansas City Cardiomyopathy Questionnaire -Total Symptom Score change from baseline at 48 weeks: number analyzed (Participants) | 194 | 204 | 193
  Kansas City Cardiomyopathy Questionnaire -Total Symptom Score change from baseline at 48 weeks | 12.78 [10.25 to 15.30] | 11.98 [9.50 to 14.46] | 13.03 [10.47 to 15.58]
Statistical Analysis 1: Comparison: AZD4831 2.5 mg vs Placebo; Change from baseline at 24 weeks; Test type: Superiority; p = 0.289, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.65, 95% CI 2-sided [-4.71 to 1.41] — Difference in adjusted mean change from baseline between AZD4831 and placebo
Statistical Analysis 2: Comparison: AZD4831 5 mg vs Placebo; Change from baseline at 24 weeks; Test type: Superiority; p = 0.571, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-3.86 to 2.13] — Difference in adjusted mean change from baseline between AZD4831 and placebo
Statistical Analysis 3: Comparison: AZD4831 2.5 mg vs Placebo; Change from baseline at 48 weeks; Test type: Superiority; p = 0.890, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-3.80 to 3.30] — Difference in adjusted mean change from baseline between AZD4831 and placebo
Statistical Analysis 4: Comparison: AZD4831 5 mg vs Placebo; Change from baseline at 48 weeks; Test type: Superiority; p = 0.558, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.04, 95% CI 2-sided [-4.55 to 2.46] — Difference in adjusted mean change from baseline between AZD4831 and placebo

4. Secondary Outcome: Six Minute Walk Distance
Description: Six Minute Walk Distance change from baseline at 24 and 48 weeks compared with placebo Part A
Time Frame: Baseline - 24 and 48 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Meters
Arm/Group | AZD4831 2.5 mg | AZD4831 5 mg | Placebo
Number analyzed (Participants) | 234 | 240 | 235
Meters
  Six Minute Walk Distance change from baseline at 24 weeks: number analyzed (Participants) | 202 | 222 | 211
  Six Minute Walk Distance change from baseline at 24 weeks | 13.5 [7.1 to 19.8] | 18.5 [12.4 to 24.6] | 15.7 [9.4 to 22.0]
  Six Minute Walk Distance change from baseline at 48 weeks: number analyzed (Participants) | 190 | 205 | 201
  Six Minute Walk Distance change from baseline at 48 weeks | 19.2 [11.9 to 26.4] | 15.7 [8.6 to 22.7] | 13.5 [6.3 to 20.6]
Statistical Analysis 1: Comparison: AZD4831 2.5 mg vs Placebo; Change from baseline at 24 weeks; Test type: Superiority; p = 0.619, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-11.1 to 6.6] — Difference in adjusted mean change from baseline between AZD4831 and placebo
Statistical Analysis 2: Comparison: AZD4831 5 mg vs Placebo; Change from baseline at 24 weeks; Test type: Superiority; p = 0.522, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [-5.8 to 11.4] — Difference in adjusted mean change from baseline between AZD4831 and placebo
Statistical Analysis 3: Comparison: AZD4831 2.5 mg vs Placebo; Change from baseline at 48 weeks; Test type: Superiority; p = 0.267, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 5.7, 95% CI 2-sided [-4.4 to 15.8] — Difference in adjusted mean change from baseline between AZD4831 and placebo
Statistical Analysis 4: Comparison: AZD4831 5 mg vs Placebo; Change from baseline at 48 weeks; Test type: Superiority; p = 0.657, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.2, 95% CI 2-sided [-7.6 to 12.1] — Difference in adjusted mean change from baseline between AZD4831 and placebo

5. Secondary Outcome: N-terminal Pro-brain Natriuretic Peptide (NT-proBNP)
Description: NT-proBNP change from baseline at 16, 24, and 48 weeks compared with placebo Part A
Time Frame: Baseline - 16, 24 and 48 weeks
Population: as for baseline characteristics
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/L
Arm/Group | AZD4831 2.5 mg | AZD4831 5 mg | Placebo
Number analyzed (Participants) | 234 | 240 | 235
ng/L
  NT-proBNP change from baseline at 16 weeks: number analyzed (Participants) | 212 | 223 | 220
  NT-proBNP change from baseline at 16 weeks | 1.00 [0.93 to 1.08] | 0.96 [0.90 to 1.03] | 1.05 [0.98 to 1.13]
  NT-proBNP change from baseline at 24 weeks: number analyzed (Participants) | 210 | 228 | 218
  NT-proBNP change from baseline at 24 weeks | 1.00 [0.92 to 1.07] | 1.00 [0.93 to 1.08] | 0.99 [0.92 to 1.07]
  NT-proBNP change from baseline at 48 weeks: number analyzed (Participants) | 195 | 212 | 201
  NT-proBNP change from baseline at 48 weeks | 1.02 [0.94 to 1.11] | 1.00 [0.93 to 1.09] | 1.08 [0.99 to 1.17]
Statistical Analysis 1: Comparison: AZD4831 2.5 mg vs Placebo; NT-proBNP change from baseline at 16 weeks; Test type: Superiority; p = 0.312, ANCOVA — Two-sided test; Treatment group, neutrophil count stratification factor and the log-transformed baseline value are included in the model as explanatory variables; Geometric mean ratio = 0.95, 95% CI 2-sided [0.86 to 1.05] — Geometric mean ratio in change from baseline between AZD4831 and placebo
Statistical Analysis 2: Comparison: AZD4831 5 mg vs Placebo; NT-proBNP change from baseline at 16 weeks; Test type: Superiority; p = 0.070, ANCOVA — Two-sided test; [statistical method as in outcome 5, analysis 1]; Geometric mean ratio = 0.91, 95% CI 2-sided [0.83 to 1.01] — Geometric mean ratio in change from baseline between AZD4831 and placebo
Statistical Analysis 3: Comparison: AZD4831 2.5 mg vs Placebo; NT-proBNP change from baseline at 24 weeks; Test type: Superiority; p = 0.911, ANCOVA — Two-sided test; [statistical method as in outcome 5, analysis 1]; Geometric mean ratio = 1.01, 95% CI 2-sided [0.91 to 1.12] — Geometric mean ratio in change from baseline between AZD4831 and placebo
Statistical Analysis 4: Comparison: AZD4831 5 mg vs Placebo; NT-proBNP change from baseline at 24 weeks; Test type: Superiority; p = 0.837, ANCOVA — Two-sided test; [statistical method as in outcome 5, analysis 1]; Geometric mean ratio = 1.01, 95% CI 2-sided [0.91 to 1.12] — Geometric mean ratio in change from baseline between AZD4831 and placebo
Statistical Analysis 5: Comparison: AZD4831 2.5 mg vs Placebo; NT-proBNP change from baseline at 48 weeks; Test type: Superiority; p = 0.370, ANCOVA — Two-sided test; [statistical method as in outcome 5, analysis 1]; Geometric mean ratio = 0.95, 95% CI 2-sided [0.84 to 1.07] — Geometric mean ratio in change from baseline between AZD4831 and placebo
Statistical Analysis 6: Comparison: AZD4831 5 mg vs Placebo; NT-proBNP change from baseline at 48 weeks; Test type: Superiority; p = 0.205, ANCOVA — Two-sided test; [statistical method as in outcome 5, analysis 1]; Geometric mean ratio = 0.93, 95% CI 2-sided [0.83 to 1.04] — Geometric mean ratio in change from baseline between AZD4831 and placebo

6. Secondary Outcome: Left Ventricular Global Longitudinal Strain (LV-GLS)
Description: LV-GLS change from baseline at 16 and 24 weeks compared with placebo Part A.
  Left ventricular global longitudinal strain (LV-GLS) is an echocardiographic measure expressing longitudinal shortening as a percentage. A negative change from baseline indicates a better outcome.
Time Frame: Baseline - 16 and 24 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage (%)
Arm/Group | AZD4831 2.5 mg | AZD4831 5 mg | Placebo
Number analyzed (Participants) | 234 | 240 | 235
Percentage (%)
  LV-GLS change from baseline at 16 weeks: number analyzed (Participants) | 109 | 121 | 117
  LV-GLS change from baseline at 16 weeks | 0.1 [-0.5 to 0.6] | -0.5 [-1.0 to 0.0] | -0.4 [-1.0 to 0.1]
  LV-GLS change from baseline at 24 weeks: number analyzed (Participants) | 114 | 132 | 121
  LV-GLS change from baseline at 24 weeks | -0.6 [-1.1 to 0.0] | -0.9 [-1.4 to -0.4] | -1.0 [-1.5 to -0.4]
Statistical Analysis 1: Comparison: AZD4831 2.5 mg vs Placebo; Change from baseline at 16 weeks; Test type: Superiority; p = 0.183, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-0.2 to 1.2] — Difference in adjusted mean change from baseline between AZD4831 and placebo
Statistical Analysis 2: Comparison: AZD4831 5 mg vs Placebo; Change from baseline at 16 weeks; Test type: Superiority; p = 0.898, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.8 to 0.7] — Difference in adjusted mean change from baseline between AZD4831 and placebo
Statistical Analysis 3: Comparison: AZD4831 2.5 mg vs Placebo; Change from baseline at 24 weeks; Test type: Superiority; p = 0.316, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.4 to 1.1] — Difference in adjusted mean change from baseline between AZD4831 and placebo
Statistical Analysis 4: Comparison: AZD4831 5 mg vs Placebo; Change from baseline at 24 weeks; Test type: Superiority; p = 0.934, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.7 to 0.8] — Difference in adjusted mean change from baseline between AZD4831 and placebo

7. Secondary Outcome: Left Atrial Volume Index (LAVI)
Description: LAVI change from baseline at 16 and 24 weeks compared with placebo Part A.
  Left atrial volume index (LAVI) is an echocardiographic measure calculated by dividing LA volume by body surface area. A negative change from baseline indicates a better outcome.
Time Frame: Baseline - 16 and 24 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/m2
Arm/Group | AZD4831 2.5 mg | AZD4831 5 mg | Placebo
Number analyzed (Participants) | 234 | 240 | 235
mL/m2
  LAVI change from baseline at 16 weeks: number analyzed (Participants) | 184 | 196 | 184
  LAVI change from baseline at 16 weeks | -0.940 [-2.373 to 0.493] | -1.894 [-3.286 to -0.502] | -1.300 [-2.743 to 0.144]
  LAVI change from baseline at 24 weeks: number analyzed (Participants) | 176 | 201 | 189
  LAVI change from baseline at 24 weeks | 1.096 [-0.626 to 2.818] | -0.376 [-1.986 to 1.235] | 0.439 [-1.236 to 2.114]
Statistical Analysis 1: Comparison: AZD4831 2.5 mg vs Placebo; Change from baseline at 16 weeks; Test type: Superiority; p = 0.725, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.360, 95% CI 2-sided [-1.647 to 2.366] — Difference in adjusted mean change from baseline between AZD4831 and placebo
Statistical Analysis 2: Comparison: AZD4831 5 mg vs Placebo; Change from baseline at 16 weeks; Test type: Superiority; p = 0.555, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.594, 95% CI 2-sided [-2.571 to 1.382] — Difference in adjusted mean change from baseline between AZD4831 and placebo
Statistical Analysis 3: Comparison: AZD4831 2.5 mg vs Placebo; Change from baseline at 24 weeks; Test type: Superiority; p = 0.586, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.657, 95% CI 2-sided [-1.710 to 3.025] — Difference in adjusted mean change from baseline between AZD4831 and placebo
Statistical Analysis 4: Comparison: AZD4831 5 mg vs Placebo; Change from baseline at 24 weeks; Test type: Superiority; p = 0.486, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.815, 95% CI 2-sided [-3.108 to 1.478] — Difference in adjusted mean change from baseline between AZD4831 and placebo

8. Secondary Outcome: Left Ventricular Mass Index (LVMI)
Description: LVMI change from baseline at 16 and 24 weeks compared with placebo Part A.
  Left ventricular mass index (LVMI) is an echocardiographic measure calculated by dividing LVM by body surface area. A negative change from baseline indicates a better outcome.
Time Frame: Baseline - 16 and 24 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: g/m2
Arm/Group | AZD4831 2.5 mg | AZD4831 5 mg | Placebo
Number analyzed (Participants) | 234 | 240 | 235
g/m2
  LVMI change from baseline at 16 weeks: number analyzed (Participants) | 200 | 208 | 204
  LVMI change from baseline at 16 weeks | 1.3 [-1.6 to 4.2] | -0.9 [-3.8 to 1.9] | 1.4 [-1.5 to 4.2]
  LVMI change from baseline at 24 weeks: number analyzed (Participants) | 197 | 213 | 202
  LVMI change from baseline at 24 weeks | 9.8 [6.0 to 13.5] | 8.3 [4.6 to 11.9] | 9.4 [5.6 to 13.1]
Statistical Analysis 1: Comparison: AZD4831 2.5 mg vs Placebo; Change from baseline at 16 weeks; Test type: Superiority; p = 0.968, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-4.1 to 3.9] — Difference in adjusted mean change from baseline between AZD4831 and placebo
Statistical Analysis 2: Comparison: AZD4831 5 mg vs Placebo; Change from baseline at 16 weeks; Test type: Superiority; p = 0.251, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-6.3 to 1.6] — Difference in adjusted mean change from baseline between AZD4831 and placebo
Statistical Analysis 3: Comparison: AZD4831 2.5 mg vs Placebo; Change from baseline at 24 weeks; Test type: Superiority; p = 0.872, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-4.8 to 5.7] — Difference in adjusted mean change from baseline between AZD4831 and placebo
Statistical Analysis 4: Comparison: AZD4831 5 mg vs Placebo; Change from baseline at 24 weeks; Test type: Superiority; p = 0.682, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-6.2 to 4.1] — No formal hypothesis testing and p-value is not adjusted for multiple comparisons

9. Secondary Outcome: Pharmacokinetics (AZD4831 Plasma Exposure)
Description: Plasma concentrations of AZD4831 summarised by timepoint and dose level Part A
Time Frame: Baseline, 4 weeks, 12 weeks, 16 weeks, 24 weeks, 48 weeks, 52 weeks
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | AZD4831 2.5 mg | AZD4831 5 mg
Number analyzed (Participants) | 231 | 238
nmol/L
  Baseline (pre-dose) | 1.02 (19.57) | 1.01 (9.38)
  4 weeks (pre-dose): number analyzed (Participants) | 225 | 236
  4 weeks (pre-dose) | 14.45 (99.26) | 26.44 (141.88)
  12 weeks (pre-dose): number analyzed (Participants) | 208 | 211
  12 weeks (pre-dose) | 13.51 (130.33) | 25.45 (161.09)
  16 weeks (pre-dose): number analyzed (Participants) | 209 | 213
  16 weeks (pre-dose) | 13.59 (126.71) | 25.31 (159.79)
  24 weeks (pre-dose): number analyzed (Participants) | 206 | 216
  24 weeks (pre-dose) | 12.87 (146.45) | 23.08 (199.18)
  48 weeks (pre-dose): number analyzed (Participants) | 193 | 205
  48 weeks (pre-dose) | 10.36 (188.55) | 21.18 (229.28)
  52 weeks (pre-dose): number analyzed (Participants) | 195 | 208
  52 weeks (pre-dose) | 1.14 (49.22) | 1.27 (74.56)

10. Secondary Outcome: High Sensitivity CRP (hsCRP)
Description: hsCRP change from baseline at 16, 24, and 48 weeks compared with placebo Part A
Time Frame: Baseline - 16, 24 and 48 weeks
Population: as for baseline characteristics
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | AZD4831 2.5 mg | AZD4831 5 mg | Placebo
Number analyzed (Participants) | 234 | 240 | 235
mg/dL
  hsCRP change from baseline at 16 weeks: number analyzed (Participants) | 210 | 224 | 218
  hsCRP change from baseline at 16 weeks | 0.940 [0.824 to 1.073] | 1.105 [0.971 to 1.257] | 0.914 [0.802 to 1.041]
  hsCRP change from baseline at 24 weeks: number analyzed (Participants) | 209 | 229 | 210
  hsCRP change from baseline at 24 weeks | 1.029 [0.907 to 1.168] | 1.101 [0.976 to 1.243] | 0.926 [0.816 to 1.051]
  hsCRP change from baseline at 48 weeks: number analyzed (Participants) | 196 | 215 | 197
  hsCRP change from baseline at 48 weeks | 1.120 [0.973 to 1.288] | 1.127 [0.985 to 1.290] | 0.972 [0.845 to 1.119]
Statistical Analysis 1: Comparison: AZD4831 2.5 mg vs Placebo; Change from baseline at 16 weeks; Test type: Superiority; p = 0.760, ANCOVA — Two-sided test; [statistical method as in outcome 5, analysis 1]; Geometric mean ratio = 1.029, 95% CI 2-sided [0.857 to 1.236] — Geometric mean ratio in change from baseline between AZD4831 and placebo
Statistical Analysis 2: Comparison: AZD4831 5 mg vs Placebo; Change from baseline at 16 weeks; Test type: Superiority; p = 0.039, ANCOVA — Two-sided test; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio = 1.209, 95% CI 2-sided [1.010 to 1.448] — Treatment group, neutrophil count stratification factor and the log-transformed baseline value are included in the model as explanatory variables
Statistical Analysis 3: Comparison: AZD4831 2.5 mg vs Placebo; Change from baseline at 24 weeks; Test type: Superiority; p = 0.241, ANCOVA — Two-sided test; [statistical method as in outcome 5, analysis 1]; Geometric mean ratio = 1.111, 95% CI 2-sided [0.931 to 1.326] — Geometric mean ratio in change from baseline between AZD4831 and placebo
Statistical Analysis 4: Comparison: AZD4831 5 mg vs Placebo; Change from baseline at 24 weeks; Test type: Superiority; p = 0.049, ANCOVA — Two-sided test; [statistical method as in outcome 5, analysis 1]; Geometric mean ratio = 1.190, 95% CI 2-sided [1.001 to 1.414] — Geometric mean ratio in change from baseline between AZD4831 and placebo
Statistical Analysis 5: Comparison: AZD4831 2.5 mg vs Placebo; Change from baseline at 48 weeks; Test type: Superiority; p = 0.158, ANCOVA — Two-sided test; [statistical method as in outcome 5, analysis 1]; Geometric mean ratio = 1.151, 95% CI 2-sided [0.946 to 1.401] — Geometric mean ratio in change from baseline between AZD4831 and placebo
Statistical Analysis 6: Comparison: AZD4831 5 mg vs Placebo; Change from baseline at 48 weeks; Test type: Superiority; p = 0.131, ANCOVA — Two-sided test; [statistical method as in outcome 5, analysis 1]; Geometric mean ratio = 1.159, 95% CI 2-sided [0.957 to 1.404] — Geometric mean ratio in change from baseline between AZD4831 and placebo

11. Secondary Outcome: Interleukin 6 (IL-6)
Description: IL-6 change from baseline at 16, 24, and 48 weeks compared with placebo Part A
Time Frame: Baseline - 16, 24 and 48 weeks
Population: as for baseline characteristics
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/L
Arm/Group | AZD4831 2.5 mg | AZD4831 5 mg | Placebo
Number analyzed (Participants) | 234 | 240 | 235
ng/L
  IL-6 change from baseline at 16 weeks: number analyzed (Participants) | 190 | 201 | 199
  IL-6 change from baseline at 16 weeks | 1.1326 [1.0261 to 1.2502] | 1.0258 [0.9316 to 1.1295] | 1.1202 [1.0170 to 1.2339]
  IL-6 change from baseline at 24 weeks: number analyzed (Participants) | 189 | 209 | 188
  IL-6 change from baseline at 24 weeks | 1.0918 [0.9934 to 1.2000] | 1.0700 [0.9777 to 1.1711] | 0.9869 [0.8975 to 1.0852]
  IL-6 change from baseline at 48 weeks: number analyzed (Participants) | 170 | 189 | 177
  IL-6 change from baseline at 48 weeks | 1.3328 [1.2134 to 1.4639] | 1.3094 [1.1972 to 1.4321] | 1.2698 [1.1574 to 1.3931]
Statistical Analysis 1: Comparison: AZD4831 2.5 mg vs Placebo; Change from baseline at 16 weeks; Test type: Superiority; p = 0.874, ANCOVA — Two-sided test; [statistical method as in outcome 5, analysis 1]; Geometric mean ratio = 1.0111, 95% CI 2-sided [0.8819 to 1.1592] — Geometric mean ratio in change from baseline between AZD4831 and placebo
Statistical Analysis 2: Comparison: AZD4831 5 mg vs Placebo; Change from baseline at 16 weeks; Test type: Superiority; p = 0.200, ANCOVA — Two-sided test; [statistical method as in outcome 5, analysis 1]; Geometric mean ratio = 0.9157, 95% CI 2-sided [0.8002 to 1.0479] — Geometric mean ratio in change from baseline between AZD4831 and placebo
Statistical Analysis 3: Comparison: AZD4831 2.5 mg vs Placebo; Change from baseline at 24 weeks; Test type: Superiority; p = 0.135, ANCOVA — Two-sided test; [statistical method as in outcome 5, analysis 1]; Geometric mean ratio = 1.1063, 95% CI 2-sided [0.9690 to 1.2631] — Geometric mean ratio in change from baseline between AZD4831 and placebo
Statistical Analysis 4: Comparison: AZD4831 5 mg vs Placebo; Change from baseline at 24 weeks; Test type: Superiority; p = 0.220, ANCOVA — Two-sided test; [statistical method as in outcome 5, analysis 1]; Geometric mean ratio = 1.0842, 95% CI 2-sided [0.9527 to 1.2339] — Geometric mean ratio in change from baseline between AZD4831 and placebo
Statistical Analysis 5: Comparison: AZD4831 2.5 mg vs Placebo; Change from baseline at 48 weeks; Test type: Superiority; p = 0.467, ANCOVA — Two-sided test; [statistical method as in outcome 5, analysis 1]; Geometric mean ratio = 1.0496, 95% CI 2-sided [0.9211 to 1.1960] — Geometric mean ratio in change from baseline between AZD4831 and placebo
Statistical Analysis 6: Comparison: AZD4831 5 mg vs Placebo; Change from baseline at 48 weeks; Test type: Superiority; p = 0.636, ANCOVA — Two-sided test; [statistical method as in outcome 5, analysis 1]; Geometric mean ratio = 1.0312, 95% CI 2-sided [0.9080 to 1.1711] — Geometric mean ratio in change from baseline between AZD4831 and placebo

12. Other Pre Specified Outcome: Adverse Events
Description: Number of participants with Adverse Events Part A
Time Frame: Baseline - 52 weeks
Population: All participants who received at least one dose of IP. Participants treated in error were accounted for in the treatment group of the treatment actually received. A participant who received any dose of the active IP was classified as in the active IP treatment group. A participant who received both doses of active IP was classified as in the highest dose treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD4831 2.5 mg | AZD4831 5 mg | Placebo
Number analyzed (Participants) | 234 | 240 | 235
Participants | 173 | 180 | 173

13. Other Pre Specified Outcome: Vital Signs
Description: Number of participants with treatment emergent vital sign abnormalities Part A
Time Frame: Baseline - 52 weeks
Population: All participants who received at least one dose of IP. Participants treated in error were accounted for in the treatment group of the treatment actually received. A participant who received any dose of the active IP was classified as in the active IP treatment group. A participant who received both doses of active IP was classified as in the highest dose treatment group. Number analyzed is the number of participants per treatment group with a baseline value and at least one post-baseline value.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD4831 2.5 mg | AZD4831 5 mg | Placebo
Number analyzed (Participants) | 233 | 240 | 234
Participants
  Diastolic blood pressure >= 90 and increase from baseline >= 10 (mmHg) | 62 | 60 | 68
  Diastolic blood pressure < 60 and decrease from baseline >= 10 (mmHg) | 32 | 42 | 33
  Pulse rate >= 100 and increase from baseline >= 20 (beats/min) | 15 | 17 | 11
  Pulse rate < 50 and decrease from baseline >= 20 (beats/min) | 2 | 6 | 8
  Systolic blood pressure >= 140 and increase from baseline >= 20 (mmHg) | 71 | 84 | 67
  Systolic blood pressure < 90 and decrease from baseline >= 20 (mmHg) | 5 | 3 | 3

14. Other Pre Specified Outcome: Clinical Laboratory (Haematology)
Description: Number of participants with outliers for clinical laboratory (chemistry) measurements Part A
Time Frame: Baseline - 52 weeks
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | AZD4831 2.5 mg | AZD4831 5 mg | Placebo
Number analyzed (Participants) | 227 | 238 | 232
Participants
  Eosinophils >= 0.7 (10^9/L) | 4 | 4 | 8
  Eosinophils >= 1.5 (10^9/L) | 0 | 0 | 0
  Hemoglobin < 100 (g/L) | 9 | 11 | 6
  Hemoglobin < 80 (g/L) | 1 | 1 | 0
  Neutrophil count < 1.5 (10^9/L) | 2 | 7 | 3
  Neutrophil count < 1.0 (10^9/L) | 0 | 1 | 0
  Leukocytes < 3.0 (10^9/L) | 3 | 5 | 6
  Leukocytes < 2.0 (10^9/L) | 0 | 1 | 0

15. Other Pre Specified Outcome: Clinical Laboratory (Chemistry)
Description: Number of participants with outliers for clinical laboratory (chemistry) measurements Part A
Time Frame: Baseline - 52 weeks
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | AZD4831 2.5 mg | AZD4831 5 mg | Placebo
Number analyzed (Participants) | 227 | 239 | 232
Participants
  ALP > 1.5x ULN | 9 | 8 | 13
  ALP > 3x ULN | 0 | 0 | 1
  ALT > 3x ULN | 5 | 2 | 3
  ALT > 5x ULN | 2 | 0 | 1
  ALT > 10x ULN | 0 | 0 | 0
  AST > 3x ULN | 3 | 3 | 4
  AST > 5x ULN | 1 | 0 | 0
  AST > 10x ULN | 0 | 0 | 0
  Creatinine >= 1.5x baseline creatinine | 15 | 10 | 14
  Creatinine >= 2x baseline creatinine | 3 | 0 | 2
  TB > 1.5x ULN | 6 | 1 | 12
  TB > 2x ULN | 1 | 1 | 2
  AST or ALT > 3x ULN | 6 | 3 | 4
  AST or ALT > 3x ULN and TB > 2x ULN | 0 | 0 | 1
  TSH >6 (mIU/L) | 19 | 25 | 18
  TSH >=10 (mIU/L) | 12 | 6 | 3
  TSH > 6 and free T4 < LLN (mIU/L) | 2 | 1 | 0
  TSH >= 10 and free T4 < LLN (mIU/L) | 2 | 0 | 0

16. Other Pre Specified Outcome: Electrocardiogram (ECG)
Description: Number of Participants With Abnormal ECG Last On-Study Value Part A
Time Frame: Baseline - 52 weeks
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | AZD4831 2.5 mg | AZD4831 5 mg | Placebo
Number analyzed (Participants) | 226 | 239 | 232
Participants
  Normal with Normal at baseline | 43 | 52 | 49
  Abnormal, not clinically significant with Normal at baseline | 17 | 19 | 14
  Abnormal, clinically significant last on-study value with Normal at baseline | 2 | 0 | 1
  Normal with Abnormal, not clinically significant at baseline | 8 | 14 | 7
  Abnormal, not clinically significant with Abnormal, not clinically significant at baseline | 132 | 135 | 137
  Abnormal, clinically significant with Abnormal, not clinically significant at baseline | 5 | 2 | 4
  Normal with Abnormal, clinically significant at baseline | 0 | 0 | 1
  Abnormal, not clinically significant with Abnormal, clinically significant at baseline | 6 | 7 | 12
  Abnormal, clinically significant with Abnormal, clinically significant at baseline | 13 | 10 | 7

ADVERSE EVENTS:
Time Frame: The on-study period (Baseline - 52 weeks). The on-study period for is calculated from the date of the first dose of IP and to the earliest date of withdrawal of consent or date of death. If withdrawal of consent or death did not occur, it is calculated from the date of the first dose of IP and to the last study visit.
Arm/Group | AZD4831 2.5 mg | AZD4831 5 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 10/234 | 3/240 | 10/235
Serious Adverse Events (participants affected / at risk) | 60/234 | 57/240 | 56/235
Other Adverse Events (participants affected / at risk) | 49/234 | 44/240 | 45/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD4831 2.5 mg (N=234) | AZD4831 5 mg (N=240) | Placebo (N=235)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 5 (6) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 3 (3) | 1 (2) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 10 (11) | 13 (16) | 13 (15)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 2 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Alcohol use (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Brachiocephalic arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Iliac artery embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 3 (4)
Peripheral embolism (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Vascular insufficiency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Mitral valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericarditis constrictive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Scleritis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis orbital (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Citrobacter bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Fournier's gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Klebsiella urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia moraxella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 4 (4) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Chemical burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (4) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 3 (4) | 3 (3) | 2 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD4831 2.5 mg (N=234) | AZD4831 5 mg (N=240) | Placebo (N=235)
Dizziness (Nervous system disorders) | 18 (21) | 10 (12) | 12 (15)
Cardiac failure (Cardiac disorders) | 11 (14) | 11 (13) | 14 (14)
Covid-19 (Infections and infestations) | 16 (16) | 18 (18) | 15 (15)
Nasopharyngitis (Infections and infestations) | 9 (12) | 13 (15) | 15 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/02/NCT04986202/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT04986202/SAP_003.pdf